CLINICAL TRIAL: NCT01743365
Title: A Phase II, Single-arm Clinical Trial of Administration of Cisplatin and 5- Fluorouracil With Afatinib as First-line Therapy in Patients With Inoperable Gastric or Gastroesophageal Junction Cancer
Brief Title: Clinical Trial of Chemotherapy Combination Cisplatin-Fluorouracil-Afatinib in Patients With Inoperable Gastric Cancer
Acronym: A-GAPP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hellenic Cooperative Oncology Group (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HE7/12; 2011-006198-25 (EudraCT Number)
Record Dates: First submitted 2012-11-28; First posted 2012-12-06 (Estimated); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Gastric Cancer; Gastroesophageal Junction Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cisplatin-5FU-Afatinib (Experimental): Cisplatin 75mg/m2 iv administered on Day 1, 5FU 750mg/m2 at 24-hour iv infusion on Days 1-4, Afatinib (BIBW-2992) 40mg per os on Days 3-5, 8-12, 15-19 of each cycle. Administration of Afatinib will start on Day 3 of each cycle with an administration interval on each weekend ("Weekday on, Weekend off") for 21 days. The administration of the combination Cisplatin-5FU-Afatinib will be continued until disease progression, appearance of significant toxicity, completion of 6 cycles, or withdrawal of consent. At completion of 6 cycles of the combination, in the absence of disease progression, the administration of Afatinib as maintenance monotherapy will be continued until disease progression, appearance of significant toxicity, or withdrawal of consent at the weekday on-weekend off schedule.
  Interventions: Drug: Cisplatin-5FU-Afatinib

INTERVENTIONS:
Drug: Cisplatin-5FU-Afatinib

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of the combination of Cisplatin,5-Fluorouracil(5FU) and Afatinib as first-line therapy in patients with advanced gastric or gastroesophageal junction cancer. The study will include 55 patients in all. The patients will receive open-label Cisplatin intravenous 75mg/m2 on Day 1, 5FU 750mg/m2 at 24-hour intravenous infusion on Days 1-4, and Afatinib 40mg per os on Days 3-5, 8-12, 15-19.

The administration of Afatinib will start on Day 3 of each therapy cycle with an administration interval on each weekend ("Weekday on, Weekend off") for 21 days. Instructions are given on the dose reduction scheme in the presence of toxicity. The administration of the combination Cisplatin-5FU-Afatinib will be continued until disease progression, appearance of significant toxicity, completion of 6 treatment cycles, or withdrawal of consent. At completion of 6 cycles of the combination, in the absence of disease progression, the administration of Afatinib as maintenance monotherapy will be continued until disease progression, appearance of significant toxicity, or withdrawal of consent at the weekday on-weekend off schedule. Imaging will be applied once every 8 weeks, and once every 12 weeks in the Afatinib maintenance therapy phase.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histological or cytological diagnosis of gastric and/or gastroesophageal junction adenocarcinoma/carcinoma.
* Locally advanced or metastatic inoperable disease.
* Life expectancy ≥12 weeks.
* Patients who may have undergone any type of palliative treatment for localised disease, including surgical approaches and palliative radiotherapy, but not in the last four weeks before the trial.
* Adequate bone marrow, hepatic and renal functional reserves (ANC≥1500mm3, PLT≥100mm3, GFR≥50ml/min by Gault Formula, bilirubin <1.5x, Aspartate Aminotransferase (AST)/Alanine Aminotransferase (ALT) <2.5x upper normal limit or 5x in the presence of hepatic metastases).
* Patients must be able to swallow pharmaceutical tablets and to be eligible to receive intravenous chemotherapy.
* Men or women patients must be at least 18 years old.
* Performance Status Scale 0 or 1 (ECOG).
* Measurable disease according to RECIST 1.1.
* Left ventricular ejection fraction (LVEF) ≥50% (ECHO or MUGA).
* Provision of patient informed consent for participation in the study and for the use of biological material for research purposes.
* Willingness and ability to comply with scheduled medical visits, therapeutic treatment programmes, laboratory testing and other study procedures.

Exclusion Criteria:

* Previous systemic first-line therapy.
* Previous therapy with EGFR/HER Tyrosine Kinase Inhibitor (TKI) or other experimental agent.
* Diagnosis of a second malignancy, except basal cell carcinoma of the squamous epithelium or in situ carcinoma of any organ, for which an appropriate treatment has been administered without indications of relapse for 12 months.
* Presence of uncontrolled, active brain metastases (controlled brain metastases are considered those that have been irradiated and have remained stable for at least 4 weeks after radiation therapy).
* Diagnosis of spinal cord compression or carcinomatous meningitis.
* Any of the following that has occurred within 12 months before the start of the study treatment: myocardial infarction, serious or unstable angina pectoris, aortic-coronary or peripheral bypass surgery, symptomatic heart failure, vascular stroke, or transient ischemic attack, or pulmonary embolism.
* Continuing grade ≥2 heart rate abnormalities; atrial fibrillation of any grade.
* Hypertension uncontrolled by medication treatment (>150/100 mm/Hg despite the administration of best medical therapy).
* In the case of previous irradiation of locally advanced disease, absence of measurable tumor sites outside the irradiation field.
* Presence of any other disease which in the opinion of the doctor responsible constitutes a contraindication for the administration of cisplatin, 5FU or afatinib.
* Diagnosed human immunodeficiency virus (HIV) or disease associated with Acquired Immunodeficiency Syndrome (AIDS).
* Pregnancy or lactation. Female patients must be surgically sterilised, menopausal, or must consent to use effective contraception throughout the course of the trial.All female patients with reproduction ability must undergo a pregnancy test (serum or urine). The effective contraceptive technique will be determined by the main investigator or a person authorized by the investigator.
* Any other serious, acute or chronic, medical or psychiatric condition or laboratory analysis finding which, in the investigator's opinion, could create excessive danger as regards the patient's participation in the trial or administration of the trial medication may render a patient ineligible for inclusion in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2013-02-11 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2019-07-29 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. | At an average of 6 months for each patient
  Imaging will be performed once every 8 weeks during treatment with cisplatin-5FU-afatinib (6 cycles), and once every 12 weeks in the Afatinib maintenance therapy phase.

SECONDARY OUTCOMES:
Evaluation of Overall Survival (OS) | OS will be calculated from the date of treatment initiation to the date of death from any cause assessed up to 36 months.
Evaluation of Progression-Free Survival (PFS) | PFS will be calculated from the date of treatment initiation to the date of disease progression or date of death, assessed up to 36 months.
Assessment of safety and tolerability | Assessed up to 36 months
  Distribution of Adverse Events (AEs) according to severity grade.
  Evaluation of AEs will be performed:
  On Day 1 and day 10 in cycle 1,on Day 1 in cycles 2-6 (every 21 days) and on Day 1 during maintenance treatment with afatinib (every 4 weeks).
Value of prognostic and/or predictive biomarkers measured in tissue and blood samples | Tumor blocks and blood samples will be collected at baseline
  Immunochemical expression of proteins/messenger ribonucleic acid (mRNA) of the tumor that can be linked to the efficacy / safety of the treatment, the tumor angiogenesis and the mechanism of action of the combination cisplatin/5FU/Afatinib.
  In bioptic material for gastric or gastroesophageal adenocarcinoma:
  * Epidermal Growth Factor Receptor (EGFR) immunohistochemical expression;
  * EGFR gene amplification (chromosome 7 gene number by FISH);
  * mRNA levels of the EGFR ligands epiregulin and amphiregulin;
  * Kirsten Rat Sarcoma (KRAS) mutations;
  * Human Epidermal Growth Factor Receptor 2 (HER2) immunohistochemical expression and gene amplification
  * HER2 p95, Human Epidermal Growth Factor Receptor 3 (HER3), Human Epidermal Growth Factor Receptor 4 (HER4) immunohistochemical and mRNA expression
  In peripheral blood and plasma:HER2 shed extracellular domain (ECD)
  There may be additions to the biomarkers to be analysed, dependent on the clinical and bibliographical data.

CONTACTS AND LOCATIONS:
Overall Officials: George Pentheroudakis, Ass.Prof, Study Chair — Dept of Medical Oncology, Ioannina University Hospital
Locations (15):
- Greece (15):
  - 2nd Dept of Internal Medicine, Agios Savvas Cancer Hospital, Athens
  - Dept of Medical Oncology, 251 Air Force Hospital, Athens
  - 2nd Dept of Internal Medicine, General Hospital of Athens "Hippokratio", Athens
  - Oncology Section, Dept of Clinical Therapeutics, General Hospital of Athens "Alexandra", Athens
  - Division of Oncology, 2nd Dept of Internal Medicine, University Hospital "Attikon", Athens
  - 2nd Dept of Medical Oncology, Agii Anargiri Cancer Hospital, Athens
  - 3rd Dept of Medical Oncology, Agii Anargiri Cancer Hospital, Athens
  - 3rd Dept of Medical Oncology, Hygeia Hospital, Athens
  - 1st Dept of Medical Oncology, Metropolitan Hospital, Athens
  - 2nd Dept of Medical Oncology, Metropolitan Hospital, Athens
  - Dept of Medical Oncology, University Hospital of Heraklion, Heraklion
  - Dept of Medical Oncology, Ioannina University Hospital, Ioannina
  - Division of Oncology, Dept of Internal Medicine, University Hospital of Patras, Pátrai
  - Dept of Medical Oncology, Papageorgiou General Hospital, Thessaloniki
  - Dept of Medical Oncology, Thermi Clinic S.A, Thessaloniki

REFERENCES:
- [Derived] Zarkavelis G, Samantas E, Koliou GA, Papadopoulou K, Mauri D, Aravantinos G, Batistatou A, Pazarli E, Tryfonopoulos D, Tsipoura A, Bobos M, Psyrri A, Makatsoris T, Petraki C, Pectasides D, Fountzilas G, Pentheroudakis G. AGAPP: efficacy of first-line cisplatin, 5-fluorouracil with afatinib in inoperable gastric and gastroesophageal junction carcinomas. A Hellenic Cooperative Oncology Group study. Acta Oncol. 2021 Jun;60(6):785-793. doi: 10.1080/0284186X.2021.1912822. Epub 2021 May 18. PMID 34003074